CLINICAL TRIAL: NCT04846595
Title: Aspects of Vulnerability of People Living with HIV in the Alpine Arc Region
Acronym: ASPEGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-16
Record Dates: First submitted 2021-04-07; First posted 2021-04-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self questionnaire (Other): The study will be offered to all patients who have been treated for HIV infection for at least 6 months, during a follow-up consultation. A self questionnaire will be administered only once per patient during the usual consultation, there is no follow-up planned.
  Interventions: Other: self questionnaire

INTERVENTIONS:
Other: self questionnaire — Evaluate the demographic variables and medical characteristics of people living with HIV in the Alpine Arc region

SUMMARY:
HIV infection in France has become a chronic disease and treatment has allowed patients to increase their life expectancy. However, these promising results suffer from a very large variability within the socio-epidemiological subgroups, and life expectancy at 20 years of age is still one third lower than in the general population. Few studies of metropolitan cohorts investigated precariousness as an independent risk factor for mortality. The investigators chose to consider the vulnerability of people living with HIV (PLWHA) through the measurement of a validated French quantitative score, called EPICES ("Évaluation de la précarité et des inégalités de santé dans les centres d'examens de santé ", Evaluation of precariousness and health inequalities in health examination centers).

DETAILED DESCRIPTION:
HIV infection in France has become a chronic disease and treatment has allowed patients to increase their life expectancy. However, these promising results suffer from a very large variability within the socio-epidemiological subgroups, and life expectancy at 20 years of age is still one third lower than in the general population. Few studies of metropolitan cohorts investigated precariousness as an independent risk factor for mortality. The investigators chose to consider the vulnerability of people living with HIV (PLWHA) through the measurement of a validated French quantitative score, called EPICES (Evaluation of precariousness and health inequalities in health examination centers). Using a self-administered questionnaire administered during an annual follow-up visit to an infectious disease specialist, the investigators seek to define in the alpine arc region in france, socio-demographic data associated with greater precariousness among PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* Any person living with HIV presenting for consultation with their infectious disease referrer.
* Patient followed for at least 6 months for their HIV infection
* Patient with undetectable or detectable HIV viral load
* Patient of legal age at the time of the study
* Patient informed of the study and having expressed no objection to the collection of health data

Exclusion Criteria:

* Patient opposed or unable to express opposition to participation in the study
* Patient is a minor at the time of the study
* Patient taking antiretroviral therapy for less than 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Variables of vulnerability | one day
  Evaluation of the variables associated with a state of vulnerability according to the "EPICES" scale (at a threshold of 30.17/100), among the social, demographic and medical characteristics of people living with HIV in the Alpine Arc region characteristics of people living with HIV in the Alpine Arc region

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Annecy Genevois, Pringy, Haute-Savoie, France

IPD SHARING:
Plan to Share IPD: No